## **COVER PAGE**

| Official title: | The perceived | quality of li | ife in adult | t patients | with | inherited |
|---|---|---|---|---|---|---|
| ichthyosis: a | qualitative inter | rview study | | | | |

ClinicalTrials.gov ID: NCT05610306

**Document date:** 20<sup>th</sup> of November 2024

## Data analysis

All interview data were analyzed using an inductive and reflexive thematic content approach. The process involved initial coding, clustering of codes into themes and comparative analysis of the codes and (sub)categories. The initial codes were organized according to the three dimensions of the BPS-model. We derived (sub)categories grounded in the data and based on the interpretations of the researchers involved in the analysis. ATLAS.ti version 9.1.3 (Scientific Software Development GmbH) was utilized for qualitative data analysis. Data collection and analysis was stopped when data saturation was reached. Peer debriefing was conducted to review the overall coding and theme progression to increase the validity.

Supplementary Table 1. Patient demographics.

| | Patients with ichthyosis |
|---|---|
| | (N=15) |
| Male:female | 5:10 |
| Age, years, median | 53 (43–62) |
| Subtype of ichthyosis | |
| ARCI, $n/N$ | 10/15 (67) |
| EH, $n/N$ | 2/15 (13) |
| XLI, $n/N$ | 3/15 (20) |
| Co-morbidities | |
| Diabetes mellitus type $2$ , $n/N$ | 1/15 (6.7) |
| Hypertension, $n/N$ | 3/15 (20) |
| Breast cancer, $n/N$ | 1/15 (6.7) |
| Skin cancer, $n/N$ | 1/15 (6.7) |
| COPD, $n/N$ | 1/15 (6.7) |
| Marital status | |
| Unmarried, $n/N$ | 3/15 (20) |
| Married, n/N | 10/15 (67) |
| Living together, <i>n/N</i> | 2/15 (13) |
| Children, n/N | 9/15 (60) |
| Highest level of education | |
| University degree, <i>n/N</i> | 3/15 (20) |
| Higher vocational training, $n/N$ | 6/15 (40) |
| Vocational training, <i>n/N</i> | 3/15 (20) |
| Lower education, $n/N$ | 3/15 (20) |
| Work situation | |
| Fulltime, $n/N$ | 5/15 (33) |
| Part-time, $n/N$ | 6/15 (40) |
| Retired, $n/N$ | 3/15 (20) |
| Incapacitated, <i>n/N</i> | 1/15 (6.7) |
| Current treatment | , |
| Emollients, $n/N$ | 7/15 (47) |
| Urea, n/N | 3/15 (20) |
| Systemic retinoids, <i>n/N</i> | 8/15 (53) |
| Biologicals, <i>n/N</i> | 2/15 (13) |
| None or other, $n/N$ | 3/15 (20) |
| Under care of a dermatologist, n/N | 12/15 (80) |
| Member of Dutch patient association for ichthyosis, $n/N$ | 10/15 (67) |

Variables were presented as counts (percentage) and medians (interquartile range).

ARCI, autosomal recessive congenital ichthyosis. EH, epidermolytic hyperkeratosis. XLI, X-linked ichthyosis.